CLINICAL TRIAL: NCT06046898
Title: Performance of Surface Mechanomyography Using a Parasternal Patch to Measure and Detect Respiratory Drive and Effort in Healthy Volunteers - PATCH-MMG
Brief Title: Surface Mechanomyography Using a Parasternal Patch to Measure and Detect Respiratory Drive and Effort
Acronym: PATCH-MMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: Single | Purpose: Device Feasibility
Other Study IDs: 49RC22_0395
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Acute Respiratory Failure
Keywords: Acute respiratory failure; Surface mechanomyography; Respiratory effort
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Intervention Model Description: Esophageal pressure, electrical activity of the diaphram (Eadi) and sMMG will be recorded in 10 healthy subjects in spontaneous ventilation (SV) and non-invasive ventilation with or without resistance.
Who Masked: Outcomes Assessor
Masking Description: Recordings will be analysed by investigators blind to ventilation conditions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- SV - R / SV + R / PSV (Experimental): Spontaneous ventilation without resistance (SV - R) / Spontaneous ventilation with resistance (SV + R) / Pressure support ventilation (PSV)
  Interventions: Device: non-invasive ventilation with or without resistance
- SV - R / PSV / SV + R (Experimental): Spontaneous ventilation without resistance / Pressure support ventilation / Spontaneous ventilation with resistance
  Interventions: Device: non-invasive ventilation with or without resistance
- SV + R / PSV / SV - R (Experimental): Spontaneous ventilation with resistance / Pressure support ventilation / Spontaneous ventilation without resistance
  Interventions: Device: non-invasive ventilation with or without resistance
- SV + R / SV - R / PSV (Experimental): Spontaneous ventilation with resistance / Spontaneous ventilation without resistance / Pressure support ventilation
  Interventions: Device: non-invasive ventilation with or without resistance
- PSV / SV + R / SV - R (Experimental): Pressure support ventilation / Spontaneous ventilation with resistance / Spontaneous ventilation without resistance
  Interventions: Device: non-invasive ventilation with or without resistance
- PSV / SV - R / SV + R (Experimental): Pressure support ventilation / Spontaneous ventilation without resistance / Spontaneous ventilation with resistance
  Interventions: Device: non-invasive ventilation with or without resistance

INTERVENTIONS:
Device: non-invasive ventilation with or without resistance — non-invasive ventilation with or without resistance.

SUMMARY:
Surface mechanomyography (sMMG) has been proposed as a tool to study muscle mechanical activity. sMMG is a noninvasive technique using specific transducers to record muscle surface oscillations due to mechanical activity of the motor units . It could be of major interest for the detection of respiratory efforts in patients with respiratory failure. This study aims at assessing the performances of sMMG to measure and detect respiratory drive and effort in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteer
* Age > 18 and < 60
* Informed consent
* Fasting
* Subjects covered by or having the rights to medical care assurance

Exclusion Criteria:

* Obesity (BMI > 30 kg.m-2)
* Respiratory disease
* Cardiovascular disease
* Contraindication to the insertion of a nasogastric tube
* Incapacity to consent
* Pregnancy, breastfeeding
* Bad understanding of the French language,
* Other protected person according to articles L1121.7 and L1121.8 of the French Public Health Act.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Accuracy of sMMG to detect respiratory effort | 5 minutes after the beginning of recording
  Delays between the beginning of the respiratory effort detected by sMMG and Eadi and the end of the respiratory effort detected by sMMG and Eadi (msec)

SECONDARY OUTCOMES:
Comparison between sMMG-time (MMG-TP) and PTPes-Pes Peak | 5 minutes after the beginning of recording
  Accuracy of sMMG to assess the intensity of respiratory effort (in comparison with pressure-time product in cm H2O.s.min-1)
Comparison between sMMG slope & Eadi parameters | 5 minutes after the beginning of recording
  Accuracy of sMMG to assess the intensity of respiratory drive (in comparison with Eadi in microvolt)
Comparison between sMMG slope & slope Peso | 5 minutes after the beginning of recording
  Accuracy of sMMG to assess the intensity of respiratory drive (in comparison Peso in cm H20)
Delay between neural time measured by sMMG and neural time measured by Eadi | 5 minutes after the beginning of recording
  Accuracy of sMMG to assess the duration of inspiratory neural time (in comparison with Eadi in msec)

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

IPD SHARING:
Plan to Share IPD: Undecided